CLINICAL TRIAL: NCT06178913
Title: Improving Prognosis and Evaluating Patient Experience Through Exercise Intervention in Patients With Nontuberculous Mycobacterial Pulmonary Disease
Brief Title: Exercise Intervention in Patients With Nontuberculous Mycobacterial Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 4-2023-0549
Record Dates: First submitted 2023-11-22; First posted 2023-12-21 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2023-12

CONDITIONS: Nontuberculous Mycobacteria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise intervention (Experimental)
  Interventions: Other: Exercise intervention

INTERVENTIONS:
Other: Exercise intervention — The exercise intervention method is a circuit training method that combines strength training and aerobic exercise forms and consists of a total of 12 movements. Performing movements 1 to 12 in order is 1 set. After completing the set, when the heart rate returns to the plateau (less than 59% of maximum heart rate), proceed to the next set, for a total of 3 sets.

SUMMARY:
The study goal is to develop exercise intervention methods to improve the prognosis and quality of life of patients with non-tuberculous mycobacterial lung disease and to confirm the effectiveness of exercise intervention. This prospective study is scheduled to be conducted as a pre-post single-arm feasibility trial, targeting a total of 50 subjects.

DETAILED DESCRIPTION:
1. After confirming the intention to participate in the study for patients with non-tuberculous mycobacterial lung disease who meet the selection criteria, basic personal information and clinical history information are collected.
2. When three people are recruited, they are organized into one group and begin a four-week exercise program. A total of 17 groups will be recruited and 50 people will be registered, and within 1 week before and after the start of the exercise program, VO2 max, physical function (6MWT, 30s sit to stand, SPPB, Handgrip strength), Baseline PFT, Laboratory test, Quality of life test (QOL) -B, CAT) is performed.
3. Once a week for 4 weeks, full-body strength training and aerobic exercise are performed for 60 minutes with an exercise expert (supervised exercise), and the remaining 6 days a week are home-based exercises, in which the subject exercises independently at home. Write it down in participants exercise diary.
4. VO2 max, physical function (6MWT, 30s sit to stand, SPPB, handgrip strength), PFT, laboratory test, and quality of life test (QOL-B, CAT) are conducted again within one week before and after the exercise intervention is completed.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 19 to 80 years diagnosed with non-tuberculous mycobacterial lung disease according to the ATS/IDSA guideline, Patients with respiratory symptoms (cough, phlegm, difficulty breathing, etc.) at the time of selection, Patients who understand the purpose of the clinical study and voluntarily agree to participate in this clinical study

Exclusion Criteria:

Patients diagnosed with cardiovascular disease (Angina, HFrEF, arrhythmia, history of heart valve surgery, etc.), Patients who have had massive hemoptysis within the last 3 months, Patients who have difficulty moving freely due to musculoskeletal problems (osteoarthritis, intervertebral disc herniation, spinal stenosis, etc.), Patients who cannot read the consent form (e.g. illiterate, foreigner, etc.)

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
VO2max | within the first 1 week (plus or minus 1 week) after the end of exercise intervention
  The patient wears a mask that transmits inhalation and exhalation to a gas analyzer on the treadmill and a heart rate monitor that measures heart rate. The treadmill gradually increases the incline and increases the speed. When the patient runs as far as they can run and raises their hand to show the measurer, the patient's VO2max is measured by measuring the maximum amount of oxygen that can be taken in and heart rate.

SECONDARY OUTCOMES:
The 6-Minute Walk Test | within the first 1 week (plus or minus 1 week) after the end of exercise intervention
  The 6-Minute Walk Test, 30-Second Sit-to-Stand, Short Physical Performance Battery, and Muscular Strength (Handgrip strength in kilograms) are employed to assess the physical ability of our study participants.
30-Second Sit-to-Stand | within the first 1 week (plus or minus 1 week) after the end of exercise intervention
  The 6-Minute Walk Test, 30-Second Sit-to-Stand, Short Physical Performance Battery, and Muscular Strength (Handgrip strength in kilograms) are employed to assess the physical ability of our study participants.
Short Physical Performance Battery | within the first 1 week (plus or minus 1 week) after the end of exercise intervention
  The 6-Minute Walk Test, 30-Second Sit-to-Stand, Short Physical Performance Battery, and Muscular Strength (Handgrip strength in kilograms) are employed to assess the physical ability of our study participants.
Muscular strength (Handgrip strength in kilograms) | within the first 1 week (plus or minus 1 week) after the end of exercise intervention
  The 6-Minute Walk Test, 30-Second Sit-to-Stand, Short Physical Performance Battery, and Muscular Strength (Handgrip strength in kilograms) are employed to assess the physical ability of our study participants.
COPD Assessment Test | within the first 1 week (plus or minus 1 week) after the end of exercise intervention
  The COPD Assessment Test and the Quality of Life-Bronchiectasis (QOL-B) questionnaire are used for evaluating the quality of life in our study participants.
the Quality of Life-Bronchiectasis (QOL-B) questionnaire | within the first 1 week (plus or minus 1 week) after the end of exercise intervention
  The COPD Assessment Test and the Quality of Life-Bronchiectasis (QOL-B) questionnaire are used for evaluating the quality of life in our study participants.
forced vital capacity in percent | within the first 1 week (plus or minus 1 week) after the end of exercise intervention
  Forced vital capacity in percent, forced expiratory volume exhaled in the first second in percent, the forced expiratory volume in 1 s/forced vital capacity ratio in percent, and bronchodilator response in percent are utilized to evaluate lung function in our study participants.
forced expiratory volume exhaled in the first second in percent | within the first 1 week (plus or minus 1 week) after the end of exercise intervention
  Forced vital capacity in percent, forced expiratory volume exhaled in the first second in percent, the forced expiratory volume in 1 s/forced vital capacity ratio in percent, and bronchodilator response in percent are utilized to evaluate lung function in our study participants.
a forced expiratory volume in 1 s/forced vital capacity ratio in percent | within the first 1 week (plus or minus 1 week) after the end of exercise intervention
  Forced vital capacity in percent, forced expiratory volume exhaled in the first second in percent, the forced expiratory volume in 1 s/forced vital capacity ratio in percent, and bronchodilator response in percent are utilized to evaluate lung function in our study participants.
bronchodilator response in percent | within the first 1 week (plus or minus 1 week) after the end of exercise intervention
  Forced vital capacity in percent, forced expiratory volume exhaled in the first second in percent, the forced expiratory volume in 1 s/forced vital capacity ratio in percent, and bronchodilator response in percent are utilized to evaluate lung function in our study participants.
WBC count per microliter | within the first 1 week (plus or minus 1 week) after the end of exercise intervention
  WBC count per microliter, hemoglobin in grams per deciliter, albumin in grams per deciliter, and CRP in milligrams per liter are used to assess inflammation, nutrition, and anemia status in our study participants.
hemoglobin in gram per deciliter | within the first 1 week (plus or minus 1 week) after the end of exercise intervention
  WBC count per microliter, hemoglobin in grams per deciliter, albumin in grams per deciliter, and CRP in milligrams per liter are used to assess inflammation, nutrition, and anemia status in our study participants.
Albumin in gram per deciliter | within the first 1 week (plus or minus 1 week) after the end of exercise intervention
  WBC count per microliter, hemoglobin in grams per deciliter, albumin in grams per deciliter, and CRP in milligrams per liter are used to assess inflammation, nutrition, and anemia status in our study participants.
CRP in miligram per liter | within the first 1 week (plus or minus 1 week) after the end of exercise intervention
  WBC count per microliter, hemoglobin in grams per deciliter, albumin in grams per deciliter, and CRP in milligrams per liter are used to assess inflammation, nutrition, and anemia status in our study participants.
Body fat mass in kilogram | within the first 1 week (plus or minus 1 week) after the end of exercise intervention
  Body fat mass in kilograms and skeletal muscle mass in kilograms are used to assess the amount of fat and muscle in our study participants.
skeletal muscle mass in kilogram | within the first 1 week (plus or minus 1 week) after the end of exercise intervention
  Body fat mass in kilograms and skeletal muscle mass in kilograms are used to assess the amount of fat and muscle in our study participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Pulmonary and Critical Care Medicine, Department of Internal Medicine, Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No